CLINICAL TRIAL: NCT05378932
Title: Impact of Dysregulation of Core Body Temperature on Sleep in Patients With Hypohidrotic Ectodermal Dysplasia
Acronym: DEH-Somno
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP220045; 2021-A02736-35 (Other: IDRCB Number)
Record Dates: First submitted 2022-03-28; First posted 2022-05-18 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Hypohidrotic Ectodermal Dysplasia
Keywords: Hypohidrotic ectodermal dysplasia; Sleep efficiency; Circadian biological clock; Melatonin; Actigraphy; Polysomnography (PSG)
MeSH Terms: conditions — Ectodermal Dysplasia 1, Anhidrotic | interventions — Actigraphy; Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hypohidrotic ectodermal dysplasia (Experimental): Patients aged 3 to 40 years old with hypohidrotic ectodermal dysplasia.
  Interventions: Other: Actigraphy; Other: Recording of proximal and distal skin temperature and temperature of the bedroom; Other: Questionnaires assessing subjective sleep quality; Other: Sweat test; Other: Urine melatonin assay; Other: Polysomnography; Other: Standardized psychological and neuropsychological assessment
- Healthy controls (Active Comparator): Healthy controls aged 3 to 40 years old without hypohidrotic ectodermal dysplasia.
  Interventions: Other: Actigraphy; Other: Recording of proximal and distal skin temperature and temperature of the bedroom; Other: Questionnaires assessing subjective sleep quality; Other: Sweat test; Other: Urine melatonin assay; Other: Polysomnography

INTERVENTIONS:
Other: Actigraphy — Sleep efficiency recording at home by means of actigraphy during 10 consecutive days.
Other: Recording of proximal and distal skin temperature and temperature of the bedroom — Recording of proximal and distal skin temperature at home by data loggers placed on the skin during 10 consecutive days.
  Recording of temperature of the bedroom by a data logger during 10 consecutive days.
Other: Questionnaires assessing subjective sleep quality — One-off questionnaires assessing subjective sleep quality. The Pittsburgh Sleep Quality Index (PSQI) evaluates sleep quality with questions about sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medications, and daytime dysfunction during the last month.
  The Epworth Sleepiness Scale evaluates daytime sleepiness and comprises 8 items (situations) during which individuals assess how likely they would fall asleep.
Other: Sweat test — One-off measurement of sweating by a sweat test at the hospital.
Other: Urine melatonin assay — Two urine melatonin at home during 24 hours, one during a week day and one during the weekend
Other: Polysomnography — Sleep architecture assessed by a polysomnography during one night at home.
Other: Standardized psychological and neuropsychological assessment — One-off psychological and neuropsychological assessment of patients with HED during a hospital visit
  Arms: Hypohidrotic ectodermal dysplasia

SUMMARY:
The aim of the study is to compare sleep efficiency by means of actigraphy in patients with hypohidrotic ectodermal dysplasia with healthy controls.

Sleep efficiency, assessed on actigraphy, sleep architecture assessed on on polysomnography, body temperature and urine melatonin levels will be compared between the patients with hypohidrotic ectodermal dysplasia with healthy controls.

DETAILED DESCRIPTION:
Ectodermal dysplasias (ED) are rare genetic diseases characterized by a developmental abnormality of at least two of the following ectodermal derivatives: teeth, nails, pilosity and glands. In the hypohidrotic form (HED), dental abnormalities (oligodontia, hypodontia) and the decrease or even the absence of sweating are predominant. The lack of sweating, and therefore of the regulation of core body temperature, can impact the daily lives of patients as soon as the ambient temperature exceeds 23-24 ° C.

Core body temperature is one of the players of the internal biological clock that regulates sleep. Indeed, sleep is induced by a decrease in core body temperature concomitant with a peak of melatonin secretion. Consequently, the absence of sweating in HED and therefore the inability to lower core body temperature may explain the poor sleep quality reported by patients. However, sleep disturbances have not been analyzed in the literature nor the relationship between sleep quality and core body temperature in patients with HED.

The sleep of patients with HED who are followed at the national reference center for rare diseases of the skin and mucous membranes of genetic origin (MAGEC center) of the Necker-Enfants Malades hospital will be evaluated and compared to sleep of healthy controls screened within in the patient's family.

The main objective of the study is to compare the sleep efficiency evaluated on actigraphy between HED patients and healthy controls.

Sleep efficiency will be measured by means of actigraphy during 10 days and one overnight polysomnography, together with continuous recording of proximal and distal skin temperature during 10 days, one-off measurement of sweating by a sweat test and urine melatonin assay over 24 hours.

Subjective sleep quality will also be assessed by means of questionnaires in patients and healthy controls. Finally, patients with HED will also have a standardized psychological and neuropsychological assessment.

ELIGIBILITY:
Inclusion Criteria:

* Male patients with molecularly confirmed hypohidrotic ectodermal dysplasia (HED), children over 3 years of age and adults under 40 years of age. Patients will be separated into 3 age groups (3 to 6 years old, 7 to 12 years old, 13 years old and over)
* Healthy controls (control subjects), of same age group, recruited if possible within the patient's direct entourage
* Written informed consent

Exclusion Criteria:

* No social insurance
* Presence of an associated pathology known to alter the quality of sleep (neurological, cardiac, psychiatric, severe sleep apnea syndrome)
* Presence of an associated pathology causing significant psychomotor retardation, behavioral disorders with impossible cooperation or significant agitation
* Treatment with psychotropic drugs or drugs stimulating vigilance
* Patient under guardianship/curatorship

Ages: 3 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 22 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2024-01-16 (Actual)

PRIMARY OUTCOMES:
Sleep efficiency on actigraphy | 10 days
  Comparison of sleep efficiency evaluated on actigraphy between HED patients and healthy controls.
Total sleep time on actigraphy | 10 days
  Comparison of total sleep time evaluated on actigraphy between HED patients and healthy controls.
Awake after sleep onset on actigraphy | 10 days
  Comparison of wake after sleep onset evaluated on actigraphy between HED patients and healthy controls.
Sleep fragmentation index | 10 days
  Comparison of sleep fragmentation index evaluated on actigraphy between HED patients and healthy controls.

SECONDARY OUTCOMES:
Melatonin secretion cycle | 48 hours
  Comparison of the melatonin secretion cycle between DEH patients and healthy controls using the urinary quantitative assay of 6-sulfatoxymelatonin by ELISA method.
Total sleep time on polysomnography | One night
  Comparison of total sleep time evaluated on polysomnography between HED patients and healthy controls.
Sleep onset latency | One night
  Comparison of sleep onset latency evaluated on polysomnography between HED patients and healthy controls.
Sleep efficiency on polysomnography | One night
  Comparison of sleep efficiency evaluated on polysomnography between HED patients and healthy controls.
Awake after sleep onset on polysomnography | One night
  Comparison of wake after sleep onset evaluated on polysomnography between HED patients and healthy controls.
Micro-arousal index | One night
  Comparison of micro-arousal index evaluated on polysomnography between HED patients and healthy controls.
Percentage of sleep stages | One night
  Comparison of the percentage of sleep stages evaluated on polysomnography between HED patients and healthy controls.
Pittsburgh Sleep Quality Index | Day 0
  Subjective sleep quality. Pittsburgh Sleep Quality Index (PSQI) to assess sleep quality. Normal value <5.
  The Epworth Sleepiness Scale to assess daytime sleepiness (normal value <8)
Epworth Sleepiness Scale | Day 0
  Subjective sleep quality. The Epworth Sleepiness Scale to assess daytime sleepiness. Normal value <8.
  The Epworth Sleepiness Scale to assess daytime sleepiness (normal value <8)
WPPSI-IV intellectual ability test | Day 0
  Neuropsychologic tests in patients with hypohidrotic ectodermal dysplasia using the WPPSI-IV. Mean normal score is 100 ± 15. Abnormal for a score <70.
WISC-V intellectual ability tests | Day 0
  Neuropsychologic tests in patients with hypohidrotic ectodermal dysplasia using the WISC-V. Mean normal score is 100 ± 15. Abnormal for a score <70.
WAIS-IV intellectual ability tests | Day 0
  Neuropsychologic tests in patients with hypohidrotic ectodermal dysplasia using the WAIS-IV. Mean normal score is 100 ± 15. Abnormal for a score <70.
TAP attention test | Day 0
  Attention test in patients with hypohidrotic ectodermal dysplasia using the TAP test. Mean normal value of T-score is 50 ± 1. Abnormal for a T-score <30.
NEPSY-II attention test | Day 0
  Attention test in patients with hypohidrotic ectodermal dysplasia using the NEPSY-II test. Mean normal value =10 (SD3). Abnormal for a score <4).
Conners 3 attention questionnaire | Day 0
  Attention questionnaire in patients with hypohidrotic ectodermal dysplasia using Conners 3 questionnaire. Mean normal value of T-score is 50 ± 10), abnormal T-score > 69.
NEPSY-II for executive function test | Day 0
  Executive function evaluation in patients with hypohidrotic ectodermal dysplasia using the NEPSY-II Mean normal score is 10 ± 3, abnormal when score <4.
Trail Making for executive function test | Day 0
  Executive function evaluation in patients with hypohidrotic ectodermal dysplasia using the Trail Making test. Mean normal score is 10 ± 3, abnormal when score <4.
TAP subtests for executive function | Day 0
  Executive function evaluation in patients with hypohidrotic ectodermal dysplasia using the TAP subtests. Mean normal value of T-score TAP subtests is 50 ± 10, abnormal T-score is <30.
BRIEF and BRIEF-P questionnaire for executive function | Day 0
  Executive function questionnaire in patients with hypohidrotic ectodermal dysplasia using BRIEF and BRIEF-P questionnaire. Mean normal value of T-score is 50 ± 10, abnormal T-score is > 65.
Correlation between skin temperature and sleep efficiency and architecture | 10 days
  Correlation between skin temperature and sleep efficiency in patients with hypohidrotic ectodermal dysplasia and healthy controls.
  Sleep efficiency is evaluated by actigraphy results and architecture by polysomnography results.
  Skin temperature is evaluated by a data logger placed on the skin.
Correlation between skin temperature and sleep questionnaires scores | 10 days
  Correlation between skin temperature and sleep quality questionnaires scores in patients with hypohidrotic ectodermal dysplasia and healthy controls.
Correlation between skin temperature and melatonin secretion | 10 days
  Correlation between skin temperature and melatonin secretion cycle in patients with hypohidrotic ectodermal dysplasia and in control subjects.
Correlation between sleep efficiency and neuropsychological test scores | 10 days
  Correlation between sleep efficiency evaluated on actigraphy and neuropsychological test scores in patients with hypohidrotic ectodermal dysplasia.

CONTACTS AND LOCATIONS:
Overall Officials: Lucie Griffon, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Brigitte Fauroux, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris; Smail Hadj-Rabia, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No